CLINICAL TRIAL: NCT02621359
Title: A Two Week Nitazoxanidebased Quadruple Regimen for Helicobacter Pylori Therapy After Failure of Standard Triple Therapy: A Single Center Experience
Brief Title: A Two Week Nitazoxanidebased Quadruple Regimen
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Hepatology and Gastroenterology Dept., Tanta university, M.D., Principle investigator, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Quadruple therapy
Record Dates: First submitted 2015-11-27; First posted 2015-12-03 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — nitazoxanide; Levofloxacin; Ofloxacin; Doxycycline; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Quadruple therapy (Experimental): Nitazoxanide (500mg bid), Levofloxacin (500 mg once daily), Omeprazole (40 mg bid) and doxycyclin (100 mg twice daily) were prescribed for 14 days.
  Interventions: Drug: Nitazoxanide; Drug: Levofloxacin; Drug: Doxycyclin; Drug: Omeprazole

INTERVENTIONS:
Drug: Nitazoxanide — Nitazoxanide 500 mg twice daily
  Other Names: Alenia, nitclean, parazoxanide
Drug: Levofloxacin — Levofloxacin 500 mg once daily
  Other Names: Tavanic, levoxin, venaxan.
Drug: Doxycyclin — Doxycyclin 100 mg twice daily
  Other Names: Vibramycin, Doxymycin
Drug: Omeprazole — Omeprazole 40 mg twice daily
  Other Names: Omepak, Pepzole, Gasec, Risek.

SUMMARY:
Helicobacter pylori (H. pylori) infection is a global health problem as it is associated with peptic ulcers, chronic gastritis, duodenitis, and stomach cancer.

Therefore, the eradication of the pathogen is of critical importance to reduce H. pylori-related complications .

However, due to increasing antibiotic resistance, eradication of Helicobacter pylori has become more challenging. With a great decline in the eradication rate of standard triple therapy for Helicobacter pylori to below 70% in many countries.

Treatment with triple therapy, which is the most frequently recommended, fails to eradicate H. pylori in approximately 20% of cases .

DETAILED DESCRIPTION:
Designing a new rescue regimen that achieves greater than 85% eradication rate is an important target of current research.

Unfortunately, the most frequently used "rescue" or "salvage" therapy is bismuth quadruple therapy consisting of a proton pump inhibitor (PPI), tetracycline, metronidazole, and bismuth [11]. This rescue therapy is inexpensive, and relatively effective with average eradication rate of 70% when used as second-line therapy. However, disadvantages of bismuth based quadruple therapy include the large daily number of pills (sometimes exceeding 18 pills), increased dosing frequency (four times daily), and frequent side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with helicobacter infection.
* in whom the standard triple therapy (clarithromycin-based triple therapy) failed

Exclusion Criteria:

* Patients under 18 or over 65 years of age.
* Those with co-existing serious illnesses such as liver cirrhosis, uremia and gastrointestinal malignancies
* pregnancy/lactation
* having contraindication or allergy to any of the study drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with eradicated helicobacter | 1 year
  The total number of patients with eradicated helicobacter

CONTACTS AND LOCATIONS:
Overall Officials: Sherief Abd-Elsalam, lecturer, Principal Investigator — Tropical medicine-Tanta university hospital
Locations (1):
- Tropical medicine dept.-Tanta university hospital, Tanta, Egypt